CLINICAL TRIAL: NCT05612542
Title: Non-inferiority Study in Pediatric Cardiac Surgery Comparing Short 24-hour Antibiotic Prophylaxis to Extended Antibiotic Prophylaxis
Brief Title: Pediatric Cardiac Surgery Comparing Short 24-hour Antibiotic Prophylaxis to Extended Antibiotic Prophylaxis
Acronym: Prophylaxis
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7484
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Antibiotic Prophylaxis
Keywords: Antibiotic Prophylaxis; Bacterial proliferation; Bacterial infections; Postoperative infection; Pediatric cardiac surgery
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of antibiotic prophylaxis is to prevent bacterial proliferation in order to reduce the risk of postoperative infection.

Numerous recent recommendations show a benefit of a reduced duration of antibiotic prophylaxis in surgery, particularly in pediatrics.

The study focuses on the incidence of postoperative infection by comparing antibiotic prophylaxis with 2nd generation cephalosporin (G2G) for 48 hours to a short antibiotic prophylaxis protocol limited to 24 hours.

The bacterial infections considered were those said to be care-related, according to the criteria of the French Society of Anesthesia and Intensive Care if they occurred within the 3 months postoperative interval and were not present before the surgery:

* sepsis
* superficial or deep surgical site infection (mediastinitis, sternitis, scar infection)
* catheterization infection,
* urinary tract infection or
* respiratory infection such as pneumopathy acquired under mechanical ventilation

The hypothesis is that reducing the duration of antibiotic prophylaxis does not expose patients to an increased risk of infection and limits exposure to antibiotics

ELIGIBILITY:
Inclusion criteria:

* Child less than 18 years of age,
* Operated for cardiac surgery at the University Hospital of Strasbourg between January 2015 and June 2019, by sternal approach (sternotomy),
* Child and holders of parental authority who have not expressed, after information, their objections to the reuse of his for the purpose of this research.

Exclusion criteria:

* Child who has undergone thoracic heart surgery (thoracotomy),
* Child with an infection at the time of heart surgery,
* Child and parental authority holders who have expressed their objections to participating in this research

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patient, under 18 years of age, operated for cardiac surgery at the University Hospital of Strasbourg between January 2015 and June 2019, by sternal approach (sternotomy)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Number of postoperative care-related infections in cardiac surgery | 24 hours after antibiotic prophylaxis

CONTACTS AND LOCATIONS:
Locations (1):
- Service réanimation pédiatrique médico-chirurgicale spécialisée - CHU de Strasbourg - France, Strasbourg, France